CLINICAL TRIAL: NCT04318743
Title: A Bridging Trial to Compare the Pharmacokinetics of Glepaglutide (ZP1848) After Single Subcutaneous Adminstration by Vial/Syringe and by Autoinjector in Healthy Subjects
Brief Title: A Bridging Trial to Compare the PK Profile When Glepaglutide is Administered Via Vial/Syringe Versus Autoinjector.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZP1848-19045
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- autoinjector - vial/syringe - vial/syringe (Experimental): Single dose of Glepaglutide 10 mg for each treatment sequence
  Interventions: Drug: Glepaglutide
- vial/syringe - autoinjector - vial/syringe (Experimental): Single dose of Glepaglutide 10 mg for each treatment sequence
  Interventions: Drug: Glepaglutide
- vial/syringe - vial/syringe - autoinjector (Experimental): Single dose of Glepaglutide 10 mg for each treatment sequence
  Interventions: Drug: Glepaglutide

INTERVENTIONS:
Drug: Glepaglutide — GLP-2
  Other Names: ZP1848

SUMMARY:
This is an open-label, randomized, single center, 2-treatment, 3-period, 3-sequence reference-replicated, crossover trial in healthy subjects to compare the PK of glepaglutide (ZP1848) after a single SC administration by vial/syringe and by autoinjector.

DETAILED DESCRIPTION:
A total of 72 subjects will be randomized in a 1:1:1 ratio to receive 10 mg glepaglutide SC via vial/syringe (Reference) twice or autoinjector (Test) in one of the 3 treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject).
2. Healthy male or female subject aged between 18 years and 54 years, both inclusive, at screening.
3. Body mass index (BMI) >20.0 kg/m2 and <29.9 kg/m2, both inclusive, at screening.
4. Willing to maintain a stable weight for the duration of the trial.
5. In overall good health according to age (medical history, physical examination, vital signs, and laboratory assessments), as judged by the Investigator at screening.
6. Able to comply with all trial procedures.

Exclusion Criteria:

1. Significant medical history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator.
2. Subject with a history of colon cancer or a history of other cancers within the last 5 years.
3. Clinically significant abnormality from physical examination, standard 12-lead ECG, or vital signs measurements as determined by the Investigator.
4. Clinically significant abnormality in hematology, clinical chemistry, or urinalysis as determined by the Investigator (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is acceptable).
5. History of significant hypersensitivity, intolerance, suspected hypersensitivity to glepaglutide or related products, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
6. Positive results for hepatitis B surface antigens (HbsAg), hepatitis C virus (HCV) antibodies and/or human immunodeficiency virus (HIV) 1 antigen or HIV 1/2 antibodies, at screening.
7. Receipt of blood products within 2 months prior to screening.
8. Donation of blood or significant blood loss from 8 weeks prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
9. Use of any prescription medications/products (other than oral, implantable, transdermal, injectable, or intrauterine hormonal contraceptives) within 14 days prior to screening, unless deemed acceptable by the Investigator.
10. Use of any nonprescription, over-the-counter medication/products, including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations, within 7 days prior to screening unless deemed acceptable by the Investigator. Up to 2 grams per day of acetaminophen is allowed at the discretion of the Investigator.
11. Use of any medications/products known to be strong inhibitors or strong inducers of cytochrome P450 3A enzyme, including St. John's wort, within 30 days prior to screening, unless deemed acceptable by the Investigator.
12. Have previously received the investigational product.
13. Receipt of any investigational product within 60 days prior to screening. Participation in more than 3 other drug studies in the 10 months prior to screening in the current trial.
14. Previous exposure to glucagon-like peptide-1 (GLP-1), GLP-2, or analogs thereof. Previous exposure to human growth hormone, somatostatin, dipeptidyl peptidase-4 inhibitors, or analogs thereof within 6 months prior to screening.
15. Have previously completed or withdrawn from this trial or any other trial investigating glepaglutide.
16. History of alcoholism or drug/chemical abuse within 2 years prior to screening.
17. Current alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL wine).
18. Positive urine drug screen (confirmed by repeat).
19. Use of tobacco, smoking cessation products, or products containing nicotine (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine lozenges, or nicotine gum ) within 3 months prior to screening.
20. Poor peripheral venous access.
21. Positive qualitative serum pregnancy test (serum human chorionic gonadotropin) (female subjects only).
22. Female who is pregnant, breastfeeding, intends to become pregnant in the immediate future.
23. Female subject of childbearing potential who is sexually active without using adequate contraceptive methods (see Section 3.4.8) from 4 weeks prior to first admission to the clinical research center until 3 months after the last dose of trial product.*
24. Male subject, who is not surgically sterilized and sexually active with a female partner of childbearing potential, and who is not willing to use adequate contraceptive methods (see Section 3.4.8), from the first dosing until 3 months after the last dose of trial product.
25. Subjects whom, in the opinion of the Investigator, should not participate in this trial.
26. Employee of PRA or the Sponsor or otherwise dependent. * Participant is of nonchildbearing potential, if she is either surgically sterilized (ie, by tubal ligation or removal of ovaries), has undergone complete hysterectomy, or is in a menopausal state (ie, at least one year without menses and a serum follicle-stimulating hormone [FSH] >40 IU/L at screening).

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Variables | From time zero to the last time point with a measurable concentration
  Cmax = maximum concentration of ZP1848total in plasma
Pharmacokinetic Variables | from time zero to the last time point with a measurable concentration
  AUC0-t = area under the plasma ZP1848total concentration-time curve (AUC)

SECONDARY OUTCOMES:
Safety Variables | 16 weeks
  Number of subject with AE/SAE as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Stine Just Maarbjerg, PhD, Study Director — Zealand Pharma A/S
Locations (1):
- PRA Health Sciences- Location Martini, Groningen, NZ, Netherlands

IPD SHARING:
Plan to Share IPD: No